CLINICAL TRIAL: NCT04270734
Title: Neural Signatures of Processing the Temporal Features of Auditory Events: From Preterm Infancy to Adulthood
Acronym: PremaTempo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI2019_843_0041
Record Dates: First submitted 2020-02-07; First posted 2020-02-17 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Time Perception; EEG; Premature Neonates; Discrimination
Keywords: time perception; rhythm; EEG; fNIRS; ERP; premature neonates; discrimination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- normal 25-36 gestational week preterm infant (Active Comparator)
  Interventions: Procedure: EEG; Procedure: NIRS
- 25-36 gestational week preterm infant with IVH (Experimental): 25-36 gestational week preterm infant with Intraventricular haemorrhages (IVH)
  Interventions: Procedure: EEG; Procedure: NIRS

INTERVENTIONS:
Procedure: EEG — Response of the cortical network in premature aged between 25 and 36 wGA in response to auditory stimuli using High Resolution Electroencephalography will be performed
Procedure: NIRS — Response of the cortical network in premature aged between 25 and 36 wGA in response to auditory stimuli using High Density Near Infrared Spectroscopy will be performed

SUMMARY:
Premature neonates are able to discriminate phonemes and voice from 28wGA at a time the neuronal network establish contact between the environment and the cortical neurones. In the present monocentric study the investigators will analyse the response of the cortical network in premature aged between 25 and 36 wGA in response to auditory stimuli using High Resolution Electroencephalography and High Density Near Infrared Spectroscopy.

DETAILED DESCRIPTION:
Neurodevelopmental disorders may be related to functional or structural disruption of the neuronal network organization at an early stage or later in the course of development. The disruption of the initial set-up could partially explain the prevalence of neurodevelopmental risks due to prematurity. The development period between 25 and 33 wGA corresponds to the period of very great prematurity and represents a key period of neurodevelopment in terms of structural and functional establishment of neuronal networks. One way to address the functionality of the neuronal networks is to evaluate the neural response to the exogenous stimuli and to interpret the mechanisms and the developmental status of the network in their ability to develop appropriate responses.

ELIGIBILITY:
Inclusion Criteria:

* full term neonates between 25 and 36 weeks gestational age

Exclusion Criteria:

* Neonates outside the age range

Ages: 0 Days to 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
measure at which age the ability to discriminate time features occurs in premature neonates with Matlab Friedtrip toolbox | at day 0
  measure at which age the ability to discriminate time features occurs in premature neonates. For the analysis of discrimination, the investigators will use cluster analysis as implemented in the Matlab Friedtrip toolbox.

SECONDARY OUTCOMES:
variation of the ability to discriminate time features between the IVH and normal preterm groups with BESA statistical tools | at day 0
  variation of the ability to discriminate time features between the IVH and normal preterm groups. For the analysis of time-frequency responses, the investigators will use cluster randomization procedures as implemented in the BESA statistical tools.

CONTACTS AND LOCATIONS:
Overall Officials: Ghilda Ghostine, MD, Principal Investigator — CHU Amiens; Guy Kongolo, MD, Principal Investigator — CHU Amiens; Sabrina Goudjil, MD, Principal Investigator — CHU Amiens; André Léké, MD, Principal Investigator — CHU Amiens; Christèle Chazal, MD, Principal Investigator — CHU Amiens; Pierre Tourneux, Pr, Principal Investigator — CHU Amiens; Coralie Degorre, MD, Principal Investigator — CHU Amiens; Emilie Bourel, MD, Principal Investigator — CHU Amiens; Laura Routier, MD, Principal Investigator — CHU Amiens; Claire Héberlé, MD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No